CLINICAL TRIAL: NCT02427646
Title: Use of Kinematic Assessment of Hand Tremor Pre- and Post- Treatment With Botulinum Toxin Type A in Essential Tremor and Parkinson Disease
Brief Title: Kinematic-guided BoNT-A Treatment for ET and PD Tremor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Neurologist, Director of the London Movement Disorders Centre, Western University, Canada
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18445
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Tremor
Keywords: Kinematics; Botulinum toxin type A
MeSH Terms: conditions — Tremor | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ET BoNT-A treatment (Experimental): ET participants treated with kinematic-guided BoNT-A injections over 6 injection cycles
  Interventions: Drug: BoNT-A
- PD tremor BoNT-A treatment (Experimental): PD participants treated with kinematic-guided BoNT-A injections over 6 injection cycles
  Interventions: Drug: BoNT-A

INTERVENTIONS:
Drug: BoNT-A — A serotype of botulinum toxins that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction. BoNT-A peripherally applied using optimal parameters by intramuscular injections to treat tremor in the most bothersome upper extremity every 16 weeks over 96 weeks. The study will be extended for those participants who benefited and will receive treatment every 12 weeks over 96 weeks. BoNT-A dose will range from 50-300 U per arm.
  Other Names: Botulinum neurotoxin type A; IncobotulinumtoxinA

SUMMARY:
The present study attempts to fill a critical knowledge gap of BoNT A in tremor management by studying the efficacy of IncobotulinumtoxinA (Xeomin®) injection for hand tremor in essential tremor and idiopathic Parkinson disease using data regarding composition of tremor obtained through sophisticated, yet clinically accessible multi-sensor based kinematic information.

DETAILED DESCRIPTION:
Current pharmacological agents used to treat Parkinson disease (PD) tremor and essential tremor (ET) provide suboptimal benefit and are commonly associated with significant adverse effects. Botulinum toxin type A (BoNT-A) has been shown to be effective for wrist tremor though functionally bothersome muscle weakness frequently occurs. This is the longest study to date demonstrating that BoNT-A therapy coupled with kinematic guidance can provide efficacious outcomes for upper limb tremor with minimized unwanted weakness. A total of 28 PD and 24 ET participants with bothersome, disabling tremor, received six serial BoNT-A treatments every 16 weeks starting at week 0 with a follow-up visit 6 weeks following a treatment, totaling 96 weeks. Clinical scales, including Fahn-Tolosa-Marin tremor rating scale (FTM), and sensor-based tremor assessments were conducted at each visit. Kinematics was utilized to identify which arm muscles contributed to the tremulous movements and the experienced injector used clinical expertise in determining BoNT-A dosages. Following BoNT-A treatment, clinical ratings of tremor severity and functional ability (FTM) showed significant improvements following the first treatment which was maintained up to week 96 in PD and ET. Kinematics detected a significant reduction in PD and ET tremor amplitudes by 70% and 76% over the treatment course, respectively. By objectively distinguishing tremulous muscles and tremor severity, adverse effects were limited to mild perceived weakness by participants in injected muscles during follow-ups. Following the fourth treatment, BoNT-A dosages in flexor and extensor wrist muscles and biceps were reduced for those experiencing residual weakness which ultimately did not interfere with tremor relief or arm function. Kinematics is an objective method that can aid clinicians in assessing and determining optimal BoNT-A parameters to alleviate both PD and ET tremor. BoNT-A injections are tolerable and effective when focal therapy regimens are determined and optimized kinematically over a long-term

ELIGIBILITY:
Inclusion Criteria:

* Consenting male and female participants, aged 18 years to 80 years
* PD individuals diagnosed by UK Brain Bank Criteria with stage H&Y2-3 disease or ET with hand tremor in their motor dominant hand
* Stable IPD/ET medication management for the 6 month duration prior to their enrollment in the study
* Individuals with IPD will be eligible for the study only if tremor is their primary and most bothersome symptom as determined by clinical exam and patient report
* Participants who are botulinum toxin naïve for tremor management

Exclusion Criteria:

* History of stroke
* Muscle weakness or any related compartmental muscle syndrome
* Smoking
* Offending medications (Lithium, valproate, steroids, amiodarone, beta-adrenergic agonists (e.g. salbutamol))
* Contradictions per the Xeomin® drug monograph
* Patients prescribed zonisamide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2020-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, FRCPC, Principal Investigator — Clinical Neurological Sciences

REFERENCES:
- [Background] Schantz EJ, Johnson EA. Properties and use of botulinum toxin and other microbial neurotoxins in medicine. Microbiol Rev. 1992 Mar;56(1):80-99. doi: 10.1128/mr.56.1.80-99.1992. PMID 1579114
- [Background] Evidente VG, Adler CH. An update on the neurologic applications of botulinum toxins. Curr Neurol Neurosci Rep. 2010 Sep;10(5):338-44. doi: 10.1007/s11910-010-0129-z. PMID 20567945
- [Background] Benito-Leon J, Louis ED. Essential tremor: emerging views of a common disorder. Nat Clin Pract Neurol. 2006 Dec;2(12):666-78; quiz 2p following 691. doi: 10.1038/ncpneuro0347. PMID 17117170
- [Background] Pullman SL, Elibol B, Fahn S. Modulation of parkinsonian tremor by radial nerve palsy. Neurology. 1994 Oct;44(10):1861-4. doi: 10.1212/wnl.44.10.1861. PMID 7936237
- [Background] Jankovic J, Schwartz K, Clemence W, Aswad A, Mordaunt J. A randomized, double-blind, placebo-controlled study to evaluate botulinum toxin type A in essential hand tremor. Mov Disord. 1996 May;11(3):250-6. doi: 10.1002/mds.870110306. PMID 8723140
- [Background] Brin MF, Lyons KE, Doucette J, Adler CH, Caviness JN, Comella CL, Dubinsky RM, Friedman JH, Manyam BV, Matsumoto JY, Pullman SL, Rajput AH, Sethi KD, Tanner C, Koller WC. A randomized, double masked, controlled trial of botulinum toxin type A in essential hand tremor. Neurology. 2001 Jun 12;56(11):1523-8. doi: 10.1212/wnl.56.11.1523. PMID 11402109
- [Background] Wissel J, Masuhr F, Schelosky L, Ebersbach G, Poewe W. Quantitative assessment of botulinum toxin treatment in 43 patients with head tremor. Mov Disord. 1997 Sep;12(5):722-6. doi: 10.1002/mds.870120516. PMID 9380055
- [Background] Trosch RM, Pullman SL. Botulinum toxin A injections for the treatment of hand tremors. Mov Disord. 1994 Nov;9(6):601-9. doi: 10.1002/mds.870090604. PMID 7845399
- [Derived] Samotus O, Rahimi F, Lee J, Jog M. Functional Ability Improved in Essential Tremor by IncobotulinumtoxinA Injections Using Kinematically Determined Biomechanical Patterns - A New Future. PLoS One. 2016 Apr 21;11(4):e0153739. doi: 10.1371/journal.pone.0153739. eCollection 2016. PMID 27101283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol enrollment identifies participants who agreed to participate and sign the consent form (total N=54). However, in the total started participant flow, two participants did not have a high enough tremor severity or consistent tremor severity during the scripted tasks held during the kinematic technology assessment, leaving N=52 in the study
Groups:
- Essential Tremor Treatment; Parkinson Disease Tremor Treatment: IncobotulinumtoxinA: A serotype of botulinum toxins that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction. BoNT-A peripherally applied using optimal parameters by intramuscular injections to treat tremor in the most bothersome upper extremity every 16 weeks over 96 weeks. The study will be extended for those participants who benefited and will receive treatment every 12 weeks over 96 weeks. BoNT-A dose will range from 50-300 U per arm.
Period: Overall Study
Arm/Group | Essential Tremor Treatment | Parkinson Disease Tremor Treatment
Started | 24 | 28
Completed | 16 | 14
Not Completed | 8 | 14
Not completed — Lack of Efficacy | 2 | 3
Not completed — Physician Decision | 1 | 4
Not completed — Protocol Violation | 3 | 3
Not completed — Bothersome hand weakness | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Essential Tremor Treatment | Parkinson Disease Tremor Treatment | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8.9) | 65 (11.5) | 68 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 13 | 21 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 28 | 52
Number of participants receiving injection in their motor-dominant limb [Count of Participants; unit: Participants] | 16 | 27 | 43

OUTCOME MEASURES:

1. Primary Outcome: Clinical Tremor Rating Scale (Fahn-Tolosa-Marin Tremor Rating Scale)
Description: Improvement in hand tremor as determined by a reduction of >8 points on a standardized clinical assessment tool (Fahn-Tolosa-Marin Tremor Assessment Scale) pre and post Xeomin® injection using kinematic guided injection parameters for both IPD and ET. Lower scores indicate a better outcome. Means and standard deviations are provided in the data tables. FTM minimum and maximum scores range from 0 to 92 FTM points.
Time Frame: 0 to 96 weeks
Population: Mean total FTM score was compared from baseline to each time-point. Here we state the baseline and final visit scores per group
Measure: Mean (Standard Deviation); unit: scores on total FTM scale
Groups:
- Essential Tremor Treatment: IncobotulinumtoxinA: A serotype of botulinum toxins that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction. BoNT-A peripherally applied using optimal parameters by intramuscular injections to treat tremor in the most bothersome upper extremity every 16 weeks over 96 weeks. The study will be extended for those participants who benefited and will receive treatment every 12 weeks over 96 weeks. BoNT-A dose will range from 50-300 U per arm. There is reduction in the total number of participants at week 96 compared to week 0 due to lost to follow-up (change in medication and other symptoms arose (n=5), and discontinued from intervention (n=3)).
- Parkinson Disease Tremor Treatment: IncobotulinumtoxinA: A serotype of botulinum toxins that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction. BoNT-A peripherally applied using optimal parameters by intramuscular injections to treat tremor in the most bothersome upper extremity every 16 weeks over 96 weeks. The study will be extended for those participants who benefited and will receive treatment every 12 weeks over 96 weeks. BoNT-A dose will range from 50-300 U per arm. There is reduction in the total number of participants at week 96 compared to week 0 due to lost to follow-up (change in medication and other symptoms arose (n=8), and discontinued from intervention (n=6)).
Arm/Group | Essential Tremor Treatment | Parkinson Disease Tremor Treatment
Number analyzed (Participants) | 24 | 28
scores on total FTM scale
  Week 0 | 30.6 (5.5) | 19.4 (2.7)
  Week 96: number analyzed (Participants) | 16 | 14
  Week 96 | 14.9 (3.5) | 14.1 (3.4)
Statistical Analysis 1: Comparison: Essential Tremor Treatment vs Parkinson Disease Tremor Treatment; Test type: Other — A linear mixed effects (LME) model via the maximized likelihood estimation was implemented using open-source statistical software, R (version 3.3.3). The effects of each clinical and kinematic outcome measures were examined for each participant group (ET and PD arms were separately analyzed thus no interaction effects were investigated) in separate LME models ("lme4" package using "lmer" function); p < 0.05, Linear mixed effects model

2. Secondary Outcome: Kinematic Tremor Severity
Description: For two subgroups of participants: (A) those with a > 8 point improvement on the tremor rating scale and (B) those with a change ≤ 8 points on the tremor rating scale, Group A will have 50% reduction in overall tremor amplitude as measured by kinematics. Kinematic measures were graphically represented as mean angular RMS amplitude and standard deviations of the population at the wrist over three trials during scripted task. Kinematic tremor analysis is shown in angular root mean square (RMS) amplitudes
Time Frame: 96 weeks
Population: Mean kinematic tremor amplitude was compared from baseline to each time-point. Here we state the baseline and final visit tremor amplitudes per group
Measure: Mean (Standard Deviation); unit: Angular root mean square amplitude
Groups:
- ET BoNT-A Treatment: ET participants treated with kinematic-guided BoNT-A injections over 6 injection cycles. We report change in tremor severity using kinematics from week 0 to week 96.
- PD Tremor BoNT-A Treatment: PD participants treated with kinematic-guided BoNT-A injections over 6 injection cycles. We report change in tremor severity using kinematics from week 0 to week 96.
Arm/Group | ET BoNT-A Treatment | PD Tremor BoNT-A Treatment
Number analyzed (Participants) | 24 | 28
Angular root mean square amplitude
  Week 0 | 0.73 (0.69) | 1.04 (0.27)
  Week 96 | 0.15 (0.26) | 0.33 (0.11)
Statistical Analysis 1: Comparison: ET BoNT-A Treatment vs PD Tremor BoNT-A Treatment; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Linear mixed effects model; a log-transformation ofthe RMS datasets was applied for statistical analysis

ADVERSE EVENTS:
Time Frame: Any adverse event data was collected during the study conduction (0-96 weeks)
Description: Serious (life threatening) side effects with BoNT-A can happen when injections are applied to neck muscles. This study only involved upper limb injections. Although spread of toxin can cause symptoms of a serious condition called botulism.
Arm/Group | Essential Tremor Treatment | Parkinson Disease Tremor Treatment
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

LIMITATIONS AND CAVEATS:
A specialized quality of life relating to tremor in PD participants would be more appropriate due to other symptoms PD patients experience. Blinded studies are not possible as muscle weakness can be easily recognized by patients and investigators

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No